CLINICAL TRIAL: NCT01714154
Title: A Multi Center, Sequential, Open-Label, Multiple-Dose Study of Setrobuvir (STV) Alone and With Co-Administration of Ritonavir-boosted Danoprevir to Evaluate the Safety, Tolerability and Pharmacokinetics of STV, DNV, and Ritonavir (RTV) in Subjects With Mild Hepatic Impairment Compared to Healthy Controls
Brief Title: A Safety And Pharmacokinetic Study of Setrobuvir Alone and In Combination With Ritonavir-Boosted Danoprevir in Subjects With Mild Hepatic Impairment Compared to Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: NP28326; 2012-002283-28 (EudraCT Number)
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Ritonavir; setrobuvir

ARMS (2):
- A: setrobuvir (Experimental)
  Interventions: Drug: setrobuvir
- B: setrobuvir + DNV/r (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir; Drug: setrobuvir

INTERVENTIONS:
Drug: danoprevir — 100 mg orally every 12 hours
  Arms: B: setrobuvir + DNV/r
Drug: ritonavir — 100 mg orally every 12 hours
  Arms: B: setrobuvir + DNV/r
Drug: setrobuvir — 200 mg orally every 12 hours

SUMMARY:
This multi-center, fixed-sequence, open-label, multiple-dose, 2-period study will evaluate the safety, tolerability and pharmacokinetics of setrobuvir alone or in combination with ritonavir-boosted danoprevir in subjects with mild hepatic impairment compared to healthy controls. All subjects will receive multiple doses of setrobuvir orally for 10 days in Period 1 and multiple doses of setrobuvir plus ritonavir-boosted danoprevir orally for 10 days in Period 2, with a washout phase of at least 9 days between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18-65 years of age, inclusive
* Weight >/= 45.0 kg
* Body mass index (BMI) 18.0 - 35.0 kg/m2, inclusive
* Females of childbearing potential and males and their female partners of childbearing potential must agree to use two forms of non-hormonal contraception as defined by protocol
* Subjects with a history of substance abuse may be enrolled provided they have not abused drugs or alcohol for at least 6 months
* Healthy subjects only:

Medical history without major recent or ongoing pathology Laboratory values at screening and Day -1 within the normal range or showing no clinically relevant deviations

* Subjects with hepatic impairment only:

Stable mild liver disease (Child-Pugh A) of cryptogenic, post-hepatic, hepatitis B/C, or alcoholic origin Stable hepatic impairment defined as no clinically significant change in disease status within the last 30 days Must be on stable dose of medication and/or treatment regimen at least 2 weeks before dosing of study medication

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* Active infection or febrile illness </= 10 days prior to the first dose of study medication
* Uncontrolled/untreated hypertension
* Inadequate renal function
* Positive urine drug screen or positive breath alcohol test at screening and on Day -1 of each period
* An average alcohol intake of more than 2 units per day or 14 units per week until 48 hours prior to enrollment
* History of any significant drug-related allergy or hepatotoxicity
* Participation in other clinical studies with an investigational drug or new chemical entity within 3 months (6 months for biologic therapies) prior to the first dose of study medication
* Positive for HIV infection
* Any clinically significant cardiovascular or cerebrovascular disease
* Healthy subjects only:

Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, absorption of medication, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study Positive screening test for HBsAg or HCV antibody

* Subjects with hepatic impairment only:

Severe ascites at screening or Day -1 History of or current severe hepatic encephalopathy (Grade 3 or higher) Biliary liver cirrhosis or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver Positive screening test for HCV antigen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 40 days
Pharmacokinetics: Maximum plasma concentration at steady-state (Css,max) | up to 16 days
Pharmacokinetics: Total area under the concentration-time curve form time 0 to 12 hours post-dose at steady-state (AUCss,0-12h) | up to 16 days
Pharmacokinetics: Plasma concentration at steady-state 12 hours post-dose (Css, 12h) | up to 16 days

SECONDARY OUTCOMES:
Pharmacokinetics: Time to maximum plasma concentration (tmax) | up to 16 days
Pharmacokinetics: Elimination half-life (t1/2) | up to 16 days
Pharmacokinetics: Apparent oral clearance at steady-state (CLss/F) | up to 16 days
Pharmacokinetics: Cumulative amount excreted at steady-state (Aess) | up to 16 days
Pharmacokinetics: Fraction of orally administered drug excreted into urine (fe/f) | up to 16 days
Pharmacokinetics of danoprevir in combination with setrobuvir: Area under the concentration-time curve (AUC) | up to 12 days
Pharmacokinetics of ritonavir in combination with setrobuvir: Area under the concentration-time curve (AUC) | up to 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Hungary (2):
  - Balatonfüred
  - Budapest
- Warsaw, Poland